CLINICAL TRIAL: NCT04398251
Title: Department of Urology, Shanghai Xu-hui Central Hospital
Brief Title: A Randomized Clinical Trail of The Effect of Postoperative Uric Acid Control on Stone Recurrence and Renal Function in Patients With Hyperuricemia of Urolithiasis.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Xuhui Central Hospital, Shanghai (Other)
Responsible Party: Principal Investigator, Zhao Hong, Department of Urology, Xuhui Central Hospital, Shanghai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2020-043
Record Dates: First submitted 2020-05-07; First posted 2020-05-21 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Hypouricemia, Renal; Urolithiasis
Keywords: Stone prevention; Renal function; Febuxostat
MeSH Terms: conditions — Renal hypouricemia; Urolithiasis | interventions — Febuxostat

STUDY DESIGN:
Intervention Model Description: 2020.1 -2020.12 patients with urolithiasis and hyperuricemia were enrolled in the urology department of our hospital (100 cases). The patients were informed of this study before operation and randomly divided into uric acid drug control group (n = 50) and non-drug control group (n = 50).
  For non-drug control group: Patients are advised to live regularly after operation, drink plenty of water, drink more than 2000ml every day, reduce the intake of high purine food and fructose-rich beverages, increase the intake of fresh vegetables, control weight and exercise regularly.
  Uric acid drug control group:or the uric acid control group, except that lifestyle changes were the same as those in the uric acid non-drug control group, non-drug uric acid control group was given febuxostat to reduce uric acid synthesis. Febuxostat is taken at a dose of 20 mg three times a week
Masking Description: Make a random table, and the patients are divided into the group according to the random table according to the order of enrollment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Uric acid drug control group (Experimental): For the uric acid control group, except that lifestyle changes were the same as those in the uric acid non-drug control group, non-drug uric acid control group was given febuxostat to reduce uric acid synthesis. Febuxostat is taken at a dose of 40 mg three times a week
  Interventions: Drug: Febuxostat 40mg Tab
- Non-drug control group (Active Comparator): They are advised to live regularly after operation, drink plenty of water, drink more than 2000ml every day, reduce the intake of high purine food and fructose-rich beverages, increase the intake of fresh vegetables, control weight and exercise regularly.
  Interventions: Behavioral: Non-drug control group

INTERVENTIONS:
Drug: Febuxostat 40mg Tab — For the uric acid control group, except that lifestyle changes were the same as those in the uric acid non-drug control group, non-drug uric acid control group was given febuxostat to reduce uric acid synthesis. Febuxostat is taken at a dose of 40 mg three times a week.
  Arms: Uric acid drug control group
Behavioral: Non-drug control group — All patients in the group are advised to live regularly after operation, drink plenty of water, drink more than 2000ml every day, reduce the intake of high purine food and fructose-rich beverages, increase the intake of fresh vegetables, control weight and exercise regularly
  Arms: Non-drug control group

SUMMARY:
The purpose of this study was to explore the effects of uric acid control on stone recurrence and renal function in patients with calculi of hyperuricemia through a prospective controlled study.

DETAILED DESCRIPTION:
2020.1 -2020.12 patients with urolithiasis and hyperuricemia were enrolled in the urology department of our hospital (100 cases). The patients were informed of this study before operation and randomly divided into uric acid drug control group (n = 50) and non-drug control group (n = 50). The patients were followed up for 3 months, 6 months, 12 months and 18 months after operation.

Informations as age, sex, height, weight, calculation BMI, past medical history, history of gout, diabetes, hyperthyroidism, calcium supplements will be recorded.

Rapid blood glucose, serum total cholesterol, high density cholesterol, thyroid hormone detection, androgen, estrogen detection, serum sodium, potassium, chlorine, calcium, magnesium, phosphorus, serum uric acid will be tested.

Renogram test to evaluate the change of single renal function. The stones burden will be followed-up with ultrasound or kub or CT plain scan.

ELIGIBILITY:
Inclusion Criteria:

* .Over 18 years old, under 70 years old, regardless of sex .The subjects had no mental illness or language dysfunction, could understand the situation of this study and had signed an informed consent form.

.No clinical manifestations of urinary tract infection, urinary routine examination showed urinary tract infection, but urinary etiology test was negative (urinary routine leukocytosis), treated with broad-spectrum antibiotics for more than 3 days.

.Clinical manifestations of urinary tract infection, urine routine examination showed urinary tract infection, and patients with positive urinary etiology were treated with sensitive antibiotics for more than 7 days.

* Serum uric acid value ≥480 µmol / L
* urinary stones

Exclusion Criteria:

* Transplanted kidney
* Fever or urinary tract infection is not treated according to the inclusion criteria
* Pregnant women and female menstruation
* Unable to tolerate anesthesia or surgery due to severe systemic disease, heart disease, pulmonary insufficiency and important organ failure
* Patients with renal insufficiency Clcr <30 mL/min
* Those who take side effects of febuxostat，Patients with side effects of febuxostat, patients with a previous history of coronary heart disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-04-10 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Stone burdern stone burdern | Change from the base line of the stone's volume and quantity at 3 months.
  Use ultrasound or kub or CT plain scan to follow up the patients.
Stone burdern stone burdern | Change from the base line of the stone's volume and quantity at 6 months.
  Use ultrasound or kub or CT plain scan to follow up the patients.
Stone burdern stone burdern | Change from the base line of the stone's volume and quantity at 12 months.
  Use ultrasound or kub or CT plain scan to follow up the patients.
Stone burdern stone burdern | Change from the base line of the stone's volume and quantity at 18 months.
  Use ultrasound or kub or CT plain scan to follow up the patients.

SECONDARY OUTCOMES:
Renal function | Change from the base line of GFR at 6 months after the operation.
  Total and partial renal function
Renal function | Change from the base line of GFR at 12 months after the operation.
  Total and partial renal function
Renal function | Change from the base line of GFR at 18 months after the operation.
  Total and partial renal function

OTHER OUTCOMES:
Serum uric acid level | Chage from the base line at 3 months after the operation
  Serum uric acid level
Serum uric acid level | Chage from the base line at 6 months after the operation
  Serum uric acid level
Serum uric acid level | Chage from the base line at 12 months after the operation
  Serum uric acid level
Serum uric acid level | Chage from the base line at 18 months after the operation
  Serum uric acid level

CONTACTS AND LOCATIONS:
Overall Officials: JianMing Guo, PHD,M.D, Study Chair — Department of Urology, Zhongshan Hospital, Shanghai
Locations (1):
- Shanghai Xuhui Central Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
Subject information, test results